CLINICAL TRIAL: NCT05890300
Title: Effectiveness of an Occupational Back-exoskeleton on the Biomechanical Load in Manual Materials Handling - a Randomized Controlled Trial.
Brief Title: Effectiveness of an Occupational Passive Back-exoskeletons on the Biomechanical Load of Warehouse Workers.
Acronym: EXO4MMH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Collaborators: Dagrofa Logistics A/S (Unknown)
Responsible Party: Principal Investigator, Lasse Schrøder Jakobsen, Principal Investigator, Aalborg University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AAU-LBK1083
Record Dates: First submitted 2023-04-27; First posted 2023-06-06 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2024-01

CONDITIONS: Work-related Musculoskeletal Disorders
Keywords: Exoskeleton; Ergonomics; Manual materials handling

STUDY DESIGN:
Intervention Model Description: All participants will complete two test sessions: 1) a pre-test (baseline), and 2) a post-test conducted after the 24-week trial. Participants will be allocated to either an experimental group or a control group. The experimental group will conduct a 24-week intervention, while the control group will receive no intervention.
  Participants are randomized to an experimental group (EXP) or a control group (CON) stratified for age, gender, and work experience. Participants allocated to the EXP will use a passive- back exoskeleton during more than 50 % of their working hours for 24 weeks. CON will be instructed to resume their normal working routine throughout the study period. Both groups will attend weekly meetings and will fill out questionnaires every fourth week.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (INT) (Experimental): Group receiving intervention
  Interventions: Device: Use of an occupational passive back-exoskeleton
- Control (CON) (No Intervention): Group receiving no intervention

INTERVENTIONS:
Device: Use of an occupational passive back-exoskeleton — The experimental group will use an occupational passive back-exoskeleton (ShoulderX V3, Ottobock bionics) for a period of 24 weeks during working hours. The exoskeleton is designed to reduce the load of the lower back during manual materials handling. The first four weeks will serve as a familiarization period, where the workers will slowly progress in hours of exoskeleton-use, while they in the remaining twenty weeks will be free to use the exoskeleton as much as they like, with a minimum limit of 18 hours per week. The control group will carry on their normal work without any changes.
  Arms: Intervention (INT)

SUMMARY:
Development of work-related musculoskeletal disorders (WMSDs) is a common issue within logistics manual materials handling which is associated with the high physical demands of the workers. Especially back injuries are highly represented among manual workers in logistics. Occupational exoskeletons are seen as a solution to this issue, as it has shown to reduce the muscle activity during several manual handling tasks within manufacturing, construction work, mechanics, and logistics. However, there is a major gap in scientific literature on studies investigating in-field effects of exoskeleton-use on longer terms, which means that we in general have very little knowledge on the pros and cons of implementing exoskeletons in the product-line of logistics. Consequently, our current understanding of how a back-supporting occupational exoskeleton can benefit the manual workers of a logistics company is limited.

The purpose of this study is to investigate (i) the long-term effects of a passive back-exoskeleton during manual materials handling on the biomechanics of the user, (ii) the changes in comfort, well-being and productivity pre and post to implementation of passive back-exoskeleton. It is hypothesized that exoskeleton-use will maintain a reduction in muscle activity of the manual workers and increase their overall well-being without affecting their productivity.

DETAILED DESCRIPTION:
Manual materials handling (MMH) is common in warehouse work, and often includes tasks causing high physical requirements on the manual workers involved. An outcome of these strenuous tasks due to a challenging physical environment is often overexertion which can cause attrition and, in some cases, lead to sickness absences and work-related musculoskeletal disorders (WMSDs). Musculoskeletal disorders are the main cause to disabling injuries in United States businesses, leading to an annual direct cost of $14 billion. These disorders are often accompanied by low-back pain, causing the most years lived with disability worldwide. Additionally, in Denmark, 37% of all work-related disorders are related to musculoskeletal load, making it the biggest contributor to sick leave. In 2019, the annual cost of work-related injuries was estimated to USD 600 million.

Wearable personal assistive systems like exoskeletons were initially designed for rehabilitation purposes, e.g., walking aid, and later for military applications. Recently, exoskeletons have been introduced for occupational use. According to the European Agency for Safety and Health at Work (EUOSHA) body-worn exoskeletons are right now being implemented as assistive devices to manual labour at workplaces all over Europe. Occupational exoskeletons were first seen in Danish industrial companies in 2019, where it was adopted by automotive industry. Exoskeletons are an attractive solution to the issues related to the physical loads carried out by workers during MMH. Still, there is a lack of studies examining the benefits, risks, and barriers to the implementation of exoskeletons in industry. Most of the research on occupational exoskeletons have been conducted in laboratory setups or by simulating work-tasks in 'ideal' conditions, while in-situ exoskeletons use to reflect real-life aspects have almost never been investigated. Despite the lack of research, exoskeletons have been proven beneficial since lower muscle load indicated by surface electromyography and lower discomfort have been reported. Yet, several limitations because of wearing the exoskeletons have been underlined: modifications of the kinematics in form of lower range of motion and increased heart rate. Additionally, it is found that unloading of a specific joint can induce increased loading of other body areas, leading to higher fatigue and exertion, besides mixed effects on heart rate and usability.

Current research indicates that occupational exoskeletons decrease the biomechanical load during MMH. This can lead to a positive effect towards the development of muscle fatigue of target areas of the body and work-related musculoskeletal disorders. Yet, there are many unexplored aspects of the implementations of exoskeletons to occupational use regarding neuromuscular coordination, changes in kinematics, discomfort, postural strain (due to the weight of the exoskeleton) and difficulty for workers to perform smooth movement.

This underlines the need to clarify the pros and cons of occupational exoskeleton use. To improve the implementation of the exoskeletons in the industry, it is important to determinate which working tasks is suitable for which exoskeletons. Furthermore, it is relevant to identify which environmental conditions that may contraindicate the use of occupational exoskeletons, e.g., working in a confined space or the need of high physical precision. Concluding, to explore the important factors driving the adoption of occupational exoskeletons for industrial use, in particular identification of key facilitators and barriers, a large-scale of field studies is needed, before being able to identify the benefits and limitations of the implementation of exoskeleton use. Such studies should include a wide range of workers and working tasks and include health-relevant outcomes like musculoskeletal disorders.

Thus, the purpose of this study is to investigate the long-term effects of exoskeleton-use during MMH. In this study, the warehouse workers will participate in a 24-week randomized controlled trial (RCT) investigating the prospective effects of a passive back-exoskeleton-use. The exoskeleton used in the present study is based on initial findings of a 5-week trial, which showed that this exoskeleton induced higher acceptance among the workers (attendance), and lower discomfort. During the intervention, parameters of muscular and kinematic changes, perceived effort, comfort and performance, liking, exertion, musculoskeletal discomfort, and productivity will be monitored.

ELIGIBILITY:
Inclusion Criteria:

I) full-time employed at the F&G department at Dagrofa Logistics A/S. II) no major injuries affecting their daily work. III) no plans of retiring before the end of the study period.

Exclusion Criteria:

I) body compositions unable to fit the exoskeleton (bad fit). II) part-time workers. III) previous low-back injury

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-09-20 (Actual); Primary Completion 2024-05-20 (Actual); Study Completion 2024-09-20 (Actual)

PRIMARY OUTCOMES:
Biomechanics | Pre-test (baseline) initial to the 24-week randomized controlled trial, and post-test subsequent the 24-week randomized controlled trial.
  Changes in the biomechanics of the back i) with / without wearing the passive back-exoskeleton during manual handling tasks, and ii) pre / post the 24-week trial when wearing the passive back-exoskeleton during manual handling tasks. Muscle activity will be collected using surface electromyography (sEMG) of the erectus spinae, descent trapezius and rectus abdominis muscles, while kinematics will be collected using inertial measurement unit (IMU) based motion capture. In relation to previous studies conducted in the PhD (study 1 and 2), the 10th and 90th percentile of sEMG amplitude and joint angles during the work tasks will be investigated.

SECONDARY OUTCOMES:
Perceived effort | Pre-test (baseline) initial to the 24-week randomized controlled trial, and post-test subsequent the 24-week randomized controlled trial.
  assessed using Borg Category-Ratio (CR) scale (0 = No effort, 10 = Maximal effort) to evaluate the work tasks conducted during the pre- and post-tests.
Comfort and Performance | Pre-test (baseline) initial to the 24-week randomized controlled trial, and post-test subsequent the 24-week randomized controlled trial.
  assessed using a questionnaire including questions on fit and (thermal) comfort, balance, range-of-motion, safety, and perceived job performance. All questions are answered using a 10-point likert-scale (e.g., 0 = no discomfort and 10 = most discomfort) [13]. The questionnaire will be filled at baseline and every fourth week during the trial.
Liking | Pre-test (baseline) initial to the 24-week randomized controlled trial, and post-test subsequent the 24-week randomized controlled trial.
  assessed using open-ended questions on liking: Q1: "What do you most like about the exoskeleton?", Q2: "What do you least like about the exoskeleton?", Q3: "If you could change anything about the exoskeleton, what would you change?" [13]. The questions will be answered at baseline and every fourth week during the trial.
Exertion | Pre-test (baseline) initial to the 24-week randomized controlled trial, and post-test subsequent the 24-week randomized controlled trial.
  assessed using a questionnaire including questions on exertion. All question are answered using a 10-point likert-scale (e.g. 0 = strongly disagree and 10 = strongly agree) [14]. The questionnaire will be filled at baseline and every fourth week during the trial.
Musculoskeletal discomfort | Pre-test (baseline) initial to the 24-week randomized controlled trial, and post-test subsequent the 24-week randomized controlled trial.
  assessed using the Cornell Musculoskeletal Discomfort Questionnaire [15]. The questionnaire will be filled at baseline and every fourth week during the trial.
Productivity | Pre-test (baseline) initial to the 24-week randomized controlled trial, and post-test subsequent the 24-week randomized controlled trial.
  assessed using Dagrofa Logistics A/S normal measurement for productivity of the worker. Changes in productivity will be tracked on a weekly basis.

OTHER OUTCOMES:
Self-reporting of exoskeleton-use during the 24-week trial | Reported every week up to 24 weeks of the intervention
  The self-reporting will be an estimation of weekly use (in hours) of the exoskeleton.

CONTACTS AND LOCATIONS:
Overall Officials: Pascal Madeleine, Professor, Study Director — Aalborg University
Locations (1):
- Aalborg University, Gistrup, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Skals S, Blafoss R, Andersen MS, de Zee M, Andersen LL. Manual material handling in the supermarket sector. Part 1: Joint angles and muscle activity of trapezius descendens and erector spinae longissimus. Appl Ergon. 2021 Apr;92:103340. doi: 10.1016/j.apergo.2020.103340. Epub 2020 Dec 16. PMID 33340719
- [Background] Liberty Mutual Insurance. 2020. 2020 Workplace Safety Index: The Top 10 Causes of Disabling Injuries
- [Background] GBD 2017 Disease and Injury Incidence and Prevalence Collaborators. Global, regional, and national incidence, prevalence, and years lived with disability for 354 diseases and injuries for 195 countries and territories, 1990-2017: a systematic analysis for the Global Burden of Disease Study 2017. Lancet. 2018 Nov 10;392(10159):1789-1858. doi: 10.1016/S0140-6736(18)32279-7. Epub 2018 Nov 8. PMID 30496104
- [Background] Arbejdstilsynets erhvervssygdomsregister og Danmarks Statistiks Registerbaserede Arbejdsstyrke-statistik (RAS). De anmeldte erhvervssygdomme inden for branchegruppen "kontor" omfatter, ud over administrativt arbejde, også anmeldelser knyttet til fx social-og sundhedsarbejde samt omsorgs- og pædagogarbejde, hvis arbejdsgiveren er registreret som kommunal administration i stedet for fx plejehjem eller daginstitutioner.
- [Background] Arbejdsskadestatistik (2019). Arbejdsmarkedets Erhvervsforsikring.
- [Background] Peters, M. & Wischniewski, S. (2019). The impact of using exoskeletons on occupational safety and health. Federal Institute for Occupational Safety and Health.
- [Background] Ingeniøren (2019). Første exoskeletter på vej ud i danske industrivirksomheder.
- [Background] Theurel, J. & Desbrosses, K. (2019). Occupational exoskeletons: Overview of their benefits and limitations in preventing work-related musculoskeletal disorders. IISE Transactions on Occupational Ergonomics and Human Factors. Volume 7, Issue 3-4, p. 264-280.
- [Background] Theurel J, Desbrosses K, Roux T, Savescu A. Physiological consequences of using an upper limb exoskeleton during manual handling tasks. Appl Ergon. 2018 Feb;67:211-217. doi: 10.1016/j.apergo.2017.10.008. Epub 2017 Oct 16. PMID 29122192
- [Background] de Looze MP, Bosch T, Krause F, Stadler KS, O'Sullivan LW. Exoskeletons for industrial application and their potential effects on physical work load. Ergonomics. 2016 May;59(5):671-81. doi: 10.1080/00140139.2015.1081988. Epub 2015 Oct 7. PMID 26444053
- [Background] Hondzinski JM, Ikuma L, de Queiroz M, Wang C. Effects of exoskeleton use on movement kinematics during performance of common work tasks: A case study. Work. 2018;61(4):575-588. doi: 10.3233/WOR-162827. PMID 30507598
- [Background] Park JH, Kim S, Nussbaum MA, Srinivasan D. Effects of two passive back-support exoskeletons on postural balance during quiet stance and functional limits of stability. J Electromyogr Kinesiol. 2021 Apr;57:102516. doi: 10.1016/j.jelekin.2021.102516. Epub 2021 Jan 19. PMID 33493784
- [Background] Kim S, Nussbaum MA, Smets M. Usability, User Acceptance, and Health Outcomes of Arm-Support Exoskeleton Use in Automotive Assembly: An 18-month Field Study. J Occup Environ Med. 2022 Mar 1;64(3):202-211. doi: 10.1097/JOM.0000000000002438. PMID 34873132
- [Background] Kim S, Nussbaum MA, Smets M, Ranganathan S. Effects of an arm-support exoskeleton on perceived work intensity and musculoskeletal discomfort: An 18-month field study in automotive assembly. Am J Ind Med. 2021 Nov;64(11):905-914. doi: 10.1002/ajim.23282. Epub 2021 Aug 6. PMID 34363229
- [Background] Hedge, A., Morimoto, S., & McCrobie, D. (1999). Cornell musculoskeletal discomfort questionnaire. Ergonomics